CLINICAL TRIAL: NCT06099340
Title: Effects of an Eccentric Muscle Strengthening Protocol on Force Moment, Muscle Activation and Plantar Flexor Structure in Patients With Central Nervous System Injuries. A Randomized Controlled Trial in Post-stroke Patients and a Pilot Study in Spinal Cord Injured Patients.
Brief Title: Effects of an Eccentric Muscle Strengthening Protocol on Force Moment, Muscle Activation and Plantar Flexor Structure of Patients With Central Nervous System Injuries.
Acronym: RenfExc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0475
Record Dates: First submitted 2023-10-09; First posted 2023-10-25 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injured; Post-stroke
Keywords: Neurological rehabilitation; Physiotherapy; Eccentric muscle strengthening; Strength; Spastic paresis; Stroke; Spinal cord injury
MeSH Terms: conditions — Stroke; Spinal Cord Injuries

STUDY DESIGN:
Masking Description: Prospective Randomized Open Blinded End-point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental " EXC " (Experimental): eccentric strengthening + conventional rehabilitation
  Interventions: Other: muscle-strengthening program
- Comparator " CONC " (Active Comparator): concentric strengthening + conventional rehabilitation
  Interventions: Other: muscle-strengthening program

INTERVENTIONS:
Other: muscle-strengthening program — a muscle-strengthening program applied to the ankle muscles (triceps surae and dorsal flexors) in physiotherapy, as a complement to conventional rehabilitation

SUMMARY:
Neurological disorders [such as Cerebral Vascular Accident (CVA) or Spinal Cord Injury (SCI)] are among the most costly health problems to society in industrialized countries. For those affected, they generate severe restrictions in mobility, significantly altering their quality of life.

Deterioration in motor function after stroke or BM is closely linked to the level of force produced at joint level. This is influenced by adaptations (neurological and tissue) inherent to the pathophysiology of the injury, and characterized by the presence of a spastic paresis syndrome.

A great deal of effort is devoted to motor neurorehabilitation (particularly physiotherapy) in the days and weeks following neurological injury. This so-called sub-acute rehabilitation phase is designed to have a positive impact on the patient's motor recovery (to prevent the development of spastic paresis), and to prevent future severe limitations in the long term.

Disorders observed in the chronic phase (partial recovery of strength, severe orthopedic deformities) demonstrate the limits of current therapies. In view of the results obtained in healthy subjects, eccentric training now seems to be one of the most promising physiotherapy methods for recovering muscle strength and countering neurological disorders.

However, its use in the sub-acute rehabilitation phase has never been evaluated in post-stroke or post-BM patients, either in terms of its effects on the strength developed in the strengthened muscles, or more locally on the neurological and tissue disorders found in these patients in the context of spastic paresis.

The aim of this project is to evaluate the effects of an eccentric muscle-strengthening exercise protocol on neurological patients in the sub-acute phase of their neurological impairment. The protocol will be applied to the ankle joint, given its importance for walking and the significant deficits found at this level in neurological populations.We hypothesize that the strengthening protocol will improve muscle strength at the ankle, and generate beneficial adaptations to combat the spastic paresis syndrome (improved muscle activation, increased muscle length, muscle volume, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 80 years
* Patient with stroke< 6 months or Patient with spinal cord injury American Spinal Injury Association (ASIA) Impairment Scale C or D (incomplete motor impairment) < 6 months (second secondary criterion).
* Patient hospitalized for primary rehabilitation in the neurological PRM department of Nantes University Hospital.
* Patient with voluntary motricity rated between 2 and 4 on the MRC (Medical Research Council) scale

Exclusion Criteria:

History of functional surgery <3 months or intramuscular injection into plantar flexors <6 months

* Patient with osteoarticular lesions contraindicating rehabilitation
* Patient unlikely to adhere to protocol (severe cognitive impairment) and/or non-compliant
* Patient with a progressive pathology contraindicating efforts (syrinx, cancer, cardiovascular instability, etc.)
* Minors, protected adults, adults unable to give consent or pregnant women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Maximum joint force moment | 10 weeks after the start of the muscle-strengthening protocol
  The force-generating capacity of the plantar flexors will be studied by measuring the maximum joint force moment on an isokinetic ergometer

SECONDARY OUTCOMES:
Measurement of joint force moment | 14 weeks after the start of the muscle-strengthening protocol
  Measurement of joint force moment, performed on an isokinetic ergometer, in isometric condition
Measurement of joint force moment | 10 weeks after the start of the muscle-strengthening protocol
  Measurement of joint force moment, performed on an isokinetic ergometer, in isometric condition

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nantes, Nantes, France